CLINICAL TRIAL: NCT02267447
Title: Risk of Cardiovascular Disease in Canada and Burden of Health Behaviours: Development of Population-based Risk Algorithms
Brief Title: Cardiovascular Disease Population Risk Tool
Acronym: CVDPoRT
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Institute for Clinical Evaluative Sciences (Other); Statistics Canada (Unknown)
Responsible Party: Sponsor
Other Study IDs: CIHR FRN - 133550
Record Dates: First submitted 2014-10-06; First posted 2014-10-17 (Estimated); Results first posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-04

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular diseases; Clinical prediction rule; Population projection; Risk stratification; Health behavior
MeSH Terms: conditions — Cardiovascular Diseases; Health Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Derivation cohort: Eligible respondents to the combined 2001, 2003 and 2005 Canadian Community Health Surveys, conducted by Statistics Canada.
- Validation cohort: Eligible respondents to the 2007 and 2009 Canadian Community Health Surveys.

SUMMARY:
The purpose of this study is to develop, evaluate, and apply a predictive algorithm for assessing CVD risk in the community setting: the Cardiovascular Disease Population Risk Tool (CVDPoRT).

DETAILED DESCRIPTION:
This observational study will use the Ontario sample of the Canadian Community Health Survey (2001, 2003, 2005; 77,251 respondents) to assess risk factors - focusing on health behaviours (physical activity, diet, smoking, and alcohol use). Incident CVD outcomes will be assessed through linkage to administrative healthcare databases (619,886 person-years of follow-up until 31 December 2011). Socio-demographic factors (age, sex, immigrant status, education) and mediating factors such as presence of diabetes and hypertension will be included as predictors. Risk prediction models will be developed using competing risks survival analysis. The analysis plan adheres to published recommendations for the development of valid risk prediction models to limit the risk of over-fitting and improve the quality of predictions. Key considerations are fully pre-specifying the predictor variables; appropriate handling of missing data; use of flexible functions for continuous predictors; and avoiding data-driven variable selection procedures that increase the risk of type I error. The 2007 and 2009 surveys (approximately 50,000 respondents) will be used for validation. Calibration will be assessed overall and in predefined subgroups of importance to clinicians and policymakers.

ELIGIBILITY:
Inclusion Criteria:

* Respondents to the Canadian Community Health Surveys

Exclusion Criteria:

* Not eligible for Ontario's universal health insurance program
* Pregnant
* Prior history of heart disease or stroke
* Younger than age 20

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The derivation cohort will be eligible respondents to the combined 2001, 2003 and 2005 Canadian Community Health Surveys, conducted by Statistics Canada. The validation cohort will consist of respondents to the 2007 and 2009 surveys.
Sampling Method: Probability Sample
Enrollment: 104219 (Actual)
Dates: Start 2000-09; Primary Completion 2014-12 (Actual); Study Completion 2016-04 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
The final model parameters will be provided in Predictive Modelling Markup Language (PMML) and Lime questionnaire files; as well, we will provide a mock dataset. These files can be used to generate risk estimates in computer applications.

REFERENCES:
- [Derived] Manuel DG, Tuna M, Bennett C, Hennessy D, Rosella L, Sanmartin C, Tu JV, Perez R, Fisher S, Taljaard M. Development and validation of a cardiovascular disease risk-prediction model using population health surveys: the Cardiovascular Disease Population Risk Tool (CVDPoRT). CMAJ. 2018 Jul 23;190(29):E871-E882. doi: 10.1503/cmaj.170914. PMID 30037888
- [Derived] Taljaard M, Tuna M, Bennett C, Perez R, Rosella L, Tu JV, Sanmartin C, Hennessy D, Tanuseputro P, Lebenbaum M, Manuel DG. Cardiovascular Disease Population Risk Tool (CVDPoRT): predictive algorithm for assessing CVD risk in the community setting. A study protocol. BMJ Open. 2014 Oct 23;4(10):e006701. doi: 10.1136/bmjopen-2014-006701. PMID 25341454

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Derivation Cohort | Validation Cohort
Started | 77251 | 26968
Completed | 77251 | 26968
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Ontario respondents of CCHS survey cycles 1.1, 2.1, 3.1 and 4.1 (conducted in 2001, 2003, 2005 and 2007, respectively). Respondents were excluded if they were not eligible for Ontario's universal health insurance program, were pregnant, self-reported a prior history of heart disease or stroke, or were age <20 at the time of survey administration.
Groups:
- Validation Cohort: Eligible respondents to the 2007/2008 Canadian Community Health Survey.
- Total: Total of all reporting groups
Arm/Group | Derivation Cohort | Validation Cohort | Total
Number analyzed (Participants) | 77,251 | 26,968 | 104219
Age, Continuous [Median (Inter-Quartile Range); unit: years]
  Female | 48.0 [35.0 to 63.0] | 51.0 [37.0 to 64.0] | 49.5 [36.0 to 63.5]
  Male | 46.0 [35.0 to 59.0] | 48.0 [35.0 to 63.0] | 47.0 [35.0 to 61.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42185 | 14801 | 56986
  Male | 35066 | 12167 | 47233

OUTCOME MEASURES:

1. Primary Outcome: Major Cardiovascular Disease Event
Description: The primary outcome of interest was a major CVD event resulting in hospitalization or sudden death from CVD. Respondents were followed from the survey administration date until the earliest of: incident event, death due to causes other than CVD (defined as a competing risk), loss to follow-up (defined as loss of health care eligibility), or end of study (31 December 2012).
Time Frame: up to 12 years
Measure: Number; unit: Cardiovascular disease event
Units Other Than Participants: person-years
Groups:
- Validation Cohort: Eligible respondents to the 2007 /2008 Canadian Community Health Surveys.
Arm/Group | Derivation Cohort | Validation Cohort
Number analyzed (Participants) | 77251 | 26938
Number analyzed (person-years) | 687135 | 131343
Cardiovascular disease event | 3182 | 527

2. Other Pre Specified Outcome: Death Due to Causes Other Than CVD
Time Frame: up to 12 years
Measure: Number; unit: deaths
Groups:
- Validation Cohort: Eligible respondents to the 2007/2008 Canadian Community Health Surveys.
Arm/Group | Derivation Cohort | Validation Cohort
Number analyzed (Participants) | 77251 | 26968
deaths | 3538 | 979

ADVERSE EVENTS:
Description: no adverse event assessment/reporting
Arm/Group | Derivation Cohort | Validation Cohort
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No